CLINICAL TRIAL: NCT02545296
Title: HIV Point-of-Care Tests in Babies Study (BABY) - Operational Evaluation of HIV Point-of-Care Tests for Very Early Infant HIV Diagnostics in Infants Born to HIV Infected Mothers in Mbeya, Tanzania
Brief Title: HIV Point-of-Care Test Evaluation in Infants
Acronym: BABY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: German Center for Infection Research (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof Dr, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LMU-IMPH-BABY-01
Record Dates: First submitted 2015-07-08; First posted 2015-09-09 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: HIV
Keywords: In-vitro Diagnostics; paediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- In-vitro Diagnostics (Other): All infants are recruited into the same arm.
  Interventions: Other: In-vitro Diagnostics

INTERVENTIONS:
Other: In-vitro Diagnostics — Ex-vivo performed diagnostic blood based test.

SUMMARY:
HIV Point-of-Care tests in Babies Study (BABY) - Operational evaluation of HIV Point-of-Care tests for very early infant HIV diagnostics in infants born to HIV infected mothers in Mbeya, Tanzania.

DETAILED DESCRIPTION:
This in-vitro diagnostic (IVD) study in infants born to HIV infected mothers evaluates the reliability and operational feasibility of an HIV Point-of-Care (PoC) test for HIV early infant diagnosis (EID) in a public health setting at obstetric clinics in Mbeya, Tanzania.

Recruitment is planned to take place at 4 obstetric/maternity study sites in and around Mbeya over a time period of 12 months. The HIV PoC test will be validated against the Standard-of-Care diagnostic test, i.e. Dried Blood Spot (DBS) analyses.

The PoC test under investigation is the Xpert HIV-1 Qual produced by Cepheid, Sunnyvale, USA.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and informed consent of the mother for her own study participation (if applicable).
2. Voluntary and informed consent of the legal guardian of the child for participation of the child in the study.
3. Mothers/legal guardians ≥18 years of age.
4. Documented maternal HIV infection.
5. Willingness to consent to HIV testing for the child and herself (if applicable).
6. Willing to consent to active tracing including home tracing.

Exclusion Criteria:

1. Deficiency in the mother, rendering it difficult, if not impossible, for her or her infant to take part in the study or understand the information provided to her. This includes alcoholism, drug dependency as well as psychiatric illnesses, suicidal tendencies or any other inability.
2. Having delivered more than 48h ago
3. Prisoners
4. Women presenting with an emergency requiring immediate medical assistance if not resolved at study inclusion.
5. Stillbirths
6. Infant requiring emergency care or born with severe malformation.
7. If within the discretion of the investigator based on recommendation of the gynaecologist or paediatrician in charge study participation would possibly add not acceptable risk or burden to the mother or infant (e.g. significant congenital malformation, health deficiencies, very low birth weight less than 1500g)
8. Unlikely to comply with protocol as judged by the principal investigator or his designate

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 604 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Specificity of PoC HIV test | Participants are planned to be followed for the duration of 6 weeks, i.e. the time point of the current Standard of Care EID
  Specificity of the PoC HIV test
Sensitivity of PoC HIV test | Participants are planned to be followed for the duration of 6 weeks, i.e. the time point of the current Standard of Care EID
  Sensitivity of the PoC HIV test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof Dr, Study Director — Medical Centre of the University of Munich
Locations (1):
- NIMR - Mbeya Medical Research Centre, Mbeya, Tanzania

REFERENCES:
- [Derived] Sabi I, Mahiga H, Mgaya J, Geisenberger O, Kastner S, Olomi W, Saathoff E, Njovu L, Lueer C, France J, Maboko L, Ntinginya NE, Hoelscher M, Kroidl A. Accuracy and Operational Characteristics of Xpert Human Immunodeficiency Virus Point-of-Care Testing at Birth and Until Week 6 in Human Immunodeficiency Virus-exposed Neonates in Tanzania. Clin Infect Dis. 2019 Feb 1;68(4):615-622. doi: 10.1093/cid/ciy538. PMID 29961841